CLINICAL TRIAL: NCT06034340
Title: Rapid Local Anesthesia by Lidocaine Administered Using STAR Particles
Brief Title: Lidocaine Administration Using STAR Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Children's Healthcare of Atlanta (Other)
Responsible Party: Principal Investigator, Eric Felner, Professor of Pediatrics, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00002928
Record Dates: First submitted 2023-08-29; First posted 2023-09-13 (Actual); Results first posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-07

CONDITIONS: Anesthesia, Local
Keywords: STAR particles; Topical Lidocaine; Skin; Pediatrics; Adolescents
MeSH Terms: interventions — Lidocaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Lidocaine-epinephrine-tetracaine (LET) Gel After and Without STAR Particle Application (Experimental): Children, adolescents, and young adults will receive local anesthesia with lidocaine-epinephrine-tetracaine (LET) gel via different methods on different arms. One arm will have STAR particles used prior to LET gel and the other arm will have aloe gel applied prior to LET gel.
  Interventions: Device: LET Gel after STAR Particle Application (Right or Left Arm); Other: LET Gel Application without STAR Particle Application (Contralateral Arm)

INTERVENTIONS:
Device: LET Gel after STAR Particle Application (Right or Left Arm) — STAR particles are made of titanium dioxide, a widely used and safe ceramic material found in sunscreens, cosmetics, and paint. The particles vary in concentration and length in order to find the optimal concentration and length. Topical lidocaine (0.5 gm of Lidocaine in LET gel) will be applied immediately after applying a STAR particle preparation to the volar surface of the antecubital fossa.
  Other Names: STAR Particle preparation
Other: LET Gel Application without STAR Particle Application (Contralateral Arm) — Topical lidocaine (0.5 gm of Lidocaine in LET gel) will be applied immediately after applying aloe gel (control condition) to the volar surface of the antecubital fossa of the contralateral arm to the one receiving the STAR particle preparation.
  Other Names: Aloe Gel before LET Gel application; Topical Lidocaine; Control

SUMMARY:
This study is being done to answer the question: Do STAR particles (tiny pieces of ceramic with small spikes) help numbing gel (a gel that helps you feel less pain) work more quickly to provide local anesthesia or numbing in a specific area? Research participants will provide feedback on how quickly the STAR particles with the numbing gel can provide anesthesia. Participants will report their sensation at either 10 or 20 minutes after application of the numbing gel.

DETAILED DESCRIPTION:
This study aims to find out if the combination of STAR particles with numbing gel can deliver anesthesia faster than applying the gel by itself. STAR particles are very small particles with microneedles on the surface that can increase and create small punctures in the skin. The small punctures should allow for the numbing gel to work more quickly and allow the area to become numb more quickly.

After pretreatment with STAR particles (applied to the right or left arm) and aloe gel (used as a control condition in the contralateral arm) a numbing gel will be applied. A Pin-Prick test will be performed to evaluate local anesthesia from the numbing gel; half the participants will be evaluated 10 minutes after application of the numbing gel and the other half will be assessed 20 minutes after the numbing gel is applied. The study team will also assess pain after needle insertion and measure how much water is being lost from the skin using a device called a Vapometer before and after the STAR particle and aloe gel applications. Participants will have follow-up calls 24 hours and 1 week after the visit to ask about any changes to the skin where the STAR particles were applied.

ELIGIBILITY:
Inclusion Criteria:

* Children, adolescents, and young adults, 10 to 21 years of age
* In good general health as determined by a medical history
* Willing to provide informed assent with parental consent and follow study requirements

Exclusion Criteria:

* Is chronically using pain medication
* Has a plan to move to another location in the next 12 months or foresees any other reason that participation in the study would be disrupted during the next 12 months
* Has skin disorders or skin allergies
* Has any previous allergy or adverse reaction to STAR particle ingredients (Titanium Dioxide)
* Has abnormal (e.g., tattooed) skin at proposed the site(s) of STAR particle application
* Has known neurological conditions that might affect sensory function or perception of pain
* Has any condition (social or medical), which in the opinion of the investigator would make study participation unsafe, would interfere with adherence to the clinical study requirements, or would complicate data interpretation

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2023-03-19 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric I Felner, MD, MS, Principal Investigator — Emory University
Locations (1):
- Emory Children's Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tadros AR, Prausnitz MR, Felner EI. Rapid local anesthesia in children enhanced by STAR particles: a first-in-humans, randomized clinical trial. Drug Deliv Transl Res. 2026 Feb;16(2):539-548. doi: 10.1007/s13346-025-01899-5. Epub 2025 Jun 23. PMID 40549079

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Children's Healthcare of Atlanta (CHOA) at Egleston in Atlanta, Georgia, USA. Participant enrollment began March 19, 2023, and all follow-up assessments were complete by June 13, 2023.
Pre-assignment Details: All participants received local anesthesia with LET gel via different methods on different arms. One arm had STAR particles applied before LET gel and the other had aloe gel (the control condition) applied before LET gel. Assessments for sharp sensation and pain took place at 10 minutes for half (11) of the participants and at 20 minutes for the other half (11) of the participants.
Units Other Than Participants: Arms
Groups:
- LET Gel After STAR Particle Application (Right or Left Arm): STAR particles are made of titanium dioxide, a widely used and safe ceramic material found in sunscreens, cosmetics, and paint. The particles vary in concentration and length to find the optimal concentration and length. Topical lidocaine (0.5 gm of Lidocaine in LET gel) will be applied immediately after applying a STAR particle preparation to the volar surface of the antecubital fossa.
Period: Overall Study
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Started | 22; 22 Arms | 22; 22 Arms
10 Minutes After LET Gel Application | 11; 11 Arms | 11; 11 Arms
20 Minutes After LET Gel Application | 11; 11 Arms | 11; 11 Arms
Completed | 22; 22 Arms | 22; 22 Arms
Not Completed | 0; 0 Arms | 0; 0 Arms

BASELINE CHARACTERISTICS:
Population: All participants received local anesthesia with LET gel via different methods on different arms. One arm had STAR particles applied before LET gel and the opposite one had aloe gel (the control condition) applied before LET gel.
Groups:
- ALL PARTICIPANTS: All participants received local anesthesia with LETgel via different methods on different arms. One arm had STAR particles applied before LET gel and the contralateral had aloe gel (the control condition) applied before LET gel. Half of the participants (after both applications) were evaluated for sharp sensation and site pain at 10 or 20 minutes after applying the LET gel.
  STAR particles are made of titanium dioxide, a widely used and safe ceramic material found in sunscreens, cosmetics, and paint. The particles will vary in concentration and length to find the optimal concentration and length. Topical lidocaine (0.5 grams of Lidocaine in LET gel) was applied immediately after applying a STAR particle preparation to the volar surface of the antecubital fossa. For the control condition, topical lidocaine (0.5grams of Lidocaine in LET gel) was applied immediately after applying aloe gel to the volar surface of the antecubital fossa of the contralateral arm to the one receiving the STAR particle preparation.
Arm/Group | ALL PARTICIPANTS
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.36 (1.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19
  Mixed (Black/White) | 2
  Mixed (Pacific Islander/White) | 1
Region of Enrollment [Number; unit: participants]
  United States | 22
Weight [Mean (Standard Deviation); unit: kilograms (kg)] | 50.3 (13.4)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 156.7 (12.4)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 20.2 (3.8)
Body Surface Area (BSA) [Mean (Standard Deviation); unit: square meters (m^2)] | 1.47 (0.24)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Sharp (as Opposed to Dull) Sensation Over Application Area
Description: The time to achieve anesthesia is assessed as the percent of sharp (as opposed to dull) sensation reported at 10 or 20 minutes after the application of LET gel.
Time Frame: Day 1 at 10 minutes or 20 minutes after application of LET gel
Population: All 22 participants had STARS applied before the LET gel on either arm and Aloe (Control) gel was applied before the LET gel on the opposite arm. Half of the participants were assessed for sharp sensation at 10 minutes and the other half were evaluated 20 minutes after the application of LET gel in both participants' arms (STAR particle and aloe (Control) gel pretreatment).
Measure: Mean (Standard Error); unit: Percentage of area with sharp sensation
Units Other Than Participants: Arms
Groups:
- LET Gel After STAR Particle Application (Right or Left Arm): Topical lidocaine (0.5 grams of Lidocaine in LET gel) was applied immediately after applying a STAR particle preparation to the volar surface of the antecubital fossa.
- LET Gel Application Without STAR Particle Application (Contralateral Arm): Topical lidocaine (0.5 grams of Lidocaine in LET gel) was applied immediately after applying aloe gel (control condition) to the volar surface of the antecubital fossa.
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Number analyzed (Arms) | 22 | 22
Percentage of area with sharp sensation
  Assessment of the area at 10 minutes post applications: number analyzed (Participants) | 11 | 11
  Assessment of the area at 10 minutes post applications: number analyzed (Arms) | 11 | 11
  Assessment of the area at 10 minutes post applications | 51.6 (29.32) | 82.0 (18.6)
  Assessment of the area at 20 minutes post applications: number analyzed (Participants) | 11 | 11
  Assessment of the area at 20 minutes post applications: number analyzed (Arms) | 11 | 11
  Assessment of the area at 20 minutes post applications | 55.7 (21.8) | 89.0 (15.6)

2. Primary Outcome: Application Site Pain Assessment
Description: The application site pain assessment was measured by using the visual analog scale (VAS). The VAS consists of a 10 centimeter (cm) line with opposite endpoints representing "no pain" (coded as 0) and "pain as bad as it could possibly be" (coded as 10).
Time Frame: Day 1 at 10 minutes or 20 minutes after application of LET gel
Population: as for outcome 1
Measure: Mean (Standard Error); unit: score on a scale
Units Other Than Participants: Arms
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Number analyzed (Arms) | 22 | 22
score on a scale
  VAS at 10 minutes post-applications: number analyzed (Participants) | 11 | 11
  VAS at 10 minutes post-applications: number analyzed (Arms) | 11 | 11
  VAS at 10 minutes post-applications | 3.09 (1.83) | 4.09 (1.92)
  VAS at 20 minutes post-applications: number analyzed (Participants) | 11 | 11
  VAS at 20 minutes post-applications: number analyzed (Arms) | 11 | 11
  VAS at 20 minutes post-applications | 4.18 (0.96) | 5.32 (1.47)

3. Secondary Outcome: Change in Transepidermal Water Loss (TEWL)
Description: The transepidermal water loss (TEWL) was measured before and after application of the STAR particles and compared to the TEWL measurement before and after application of the aloe gel.
Time Frame: Day 1 at baseline and immediately after application of LET gel
Population: All 22 participants underwent TEWL measurements before and after the STAR and aloe (Control) gel applications.
Measure: Mean (Standard Error); unit: g/m^2/hr
Units Other Than Participants: Arms
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Number analyzed (Arms) | 22 | 22
g/m^2/hr | 25.0 (8.7) | 14.8 (4.3)

4. Secondary Outcome: Number of Participants With Acute Skin Reactions (ASRs)
Description: Participants were observed for acute skin reactions at each application site on both arms.
Time Frame: Immediately, 1 hour, 24 hours, and 7 days after application.
Measure: Count of Participants; unit: Participants
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

5. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: All adverse events were documented starting immediately after lidocaine application up to 1 week after application.
Time Frame: Immediately after application, 1 hour after application and up to 1 week after application
Measure: Count of Participants; unit: Participants
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events
Description: All serious adverse events were documented starting immediately after lidocaine application up to one week after application.
Time Frame: Immediately after application, 1 hour after application and up to 1 week after application
Measure: Count of Participants; unit: Participants
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
Number analyzed (Participants) | 22 | 22
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events, Serious Adverse Effects, and Skin changes were assessed in both arms on the day of application, 24 hours, and 7 days after completion of the study.
Arm/Group | LET Gel After STAR Particle Application (Right or Left Arm) | LET Gel Application Without STAR Particle Application (Contralateral Arm)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-04-27): https://cdn.clinicaltrials.gov/large-docs/40/NCT06034340/Prot_001.pdf